CLINICAL TRIAL: NCT02453789
Title: A Randomized Double-blind, Placebo-controlled Cross-over Study of Inhaled Alginate Oligosaccharide (OligoG) for 28 Days in Subjects With Cystic Fibrosis Using Aztreonam Due to Chronic Colonization With Burkholderia Spp.
Brief Title: A Study of OligoG in Cystic Fibrosis Subjects With Burkholderia Spp. Infection
Acronym: SMR-2591
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlgiPharma AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMR-2591
Record Dates: First submitted 2015-05-14; First posted 2015-05-27 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis; Burkholderia Infection
Keywords: alginate oligosaccharide; cystic fibrosis; Burkholderia; aztreonam
MeSH Terms: conditions — Cystic Fibrosis; Burkholderia Infections | interventions — oligoG CF-5-20

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alginate oligosaccharide (Active Comparator): Inhalation of a dry powder OligoG in the first treatment period, and placebo in the second period
  Interventions: Drug: Alginate oligosaccharide
- Placebo (Placebo Comparator): Inhalation of placebo dry powder in the first treatment period, and OligoG in the second period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alginate oligosaccharide — Inhalation of dry powder for inhalation (DPI)
  Other Names: OligoG
  Arms: Alginate oligosaccharide
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy of Alginate oligosaccharide (OligoG) dry powder for inhalation in cystic fibrosis (CF) patients with a Burkholderia spp. infection.

DETAILED DESCRIPTION:
Primary objective:

To explore the efficacy of inhaled OligoG in reducing the microbial burden of Burkholderia spp. as measured in expectorated sputum samples.

Secondary objectives:

To explore the effect of inhaled OligoG on various efficacy variables such as lung function, Quality-of-Life, rheology and other microbiological outcome measures.

To evaluate the safety, tolerability and subject compliance with treatment The study will also evaluate the effect of inhaled OligoG on various efficacy variables such as lung function, Quality-of-Life, rheology and other microbiological outcome measures, and evaluate the safety and patient compliance with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a confirmed diagnosis of cystic fibrosis defined by:

  * Clinical features consistent with the diagnosis of CF; AND
  * Sweat chloride ≥60 mmol/L by pilocarpine iontophoresis; OR
  * Genotypic confirmation of CFTR mutation
* Aged 18 years or older
* Ability to provide sputum samples for microbiological evaluation throughout the study either spontaneously or induced.
* Chronic colonization with Burkholderia spp. defined as at least two positive microbiological cultures in expectorated sputum within the last 12 months from Visit 1.
* Use of inhaled aztreonam three times daily in a 4 weeks on/off cycle treatment regimen or a continuous intake regimen for at least 4 weeks before screening visit. For on/off cycles, screening visit should take place in the off phase. Randomization visit should take place the first day "on" to harmonize the aztreonam inhalation period with the IMP intake period.
* Willingness to stop treatment with other inhaled antibiotics.
* At Screening no clinical or laboratory findings suggestive of significant pulmonary illness, other than CF, which in the opinion of the investigator would preclude participation in the study.
* FEV1 greater than 25% of the predicted normal value following adjustment for age, gender, and height according to the Global Lung Initiative
* Female subjects of child bearing potential and male subjects participating in the study who are sexually active must use acceptable contraception. Female subjects documented as being of non-child-bearing potential are exempt from the contraceptive requirements.
* Provision of written informed consent.

Exclusion Criteria:

* Changes in underlying therapy within the 14 days prior to Day 0. Subjects must be willing to remain on the same underlying stable therapy regimens for the duration of the study until the final follow-up visit at Day 98.
* Changes in physiotherapy technique or schedule within 14 days prior to Day 0.
* Prohibited medications within 7 days prior to Day 0. Concomitant administration of inhaled mannitol or hypertonic saline within 7 days prior to Day 0.
* Concomitant use of inhaled antibiotics other than aztreonam.
* Pulmonary exacerbation within 28 days of Screening.
* Lactose intolerance/milk allergy.
* On-going acute illness. Subjects must not have needed an outpatient visit, hospitalization or required any change in therapy for other pulmonary disease between Screening and Day 0.
* History of, or planned organ transplantation.
* Active allergic bronchopulmonary aspergillosis (ABPA) in the last 12 months prior to Screening, defined as having received treatment for ABPA.
* Inability or unwillingness to provide sputum samples for microbiological evaluation throughout the study either spontaneously or induced by means of using inhaled hypertonic saline.
* Clinically significant abnormal findings on haematology or clinical chemistry. In addition, any value ≥ 3 x the upper limit of normal will exclude the subject from participating in the study.
* Subjects unable to perform pulmonary function tests according to the ATS/ERS criteria.
* Pregnant or breast-feeding women. A negative urine pregnancy test must be demonstrated in females of child-bearing potential at Screening.
* Subjects who have participated in any interventional clinical trial within the 28 days prior to Day 0.
* Subjects with documented or suspected, clinically significant, alcohol or drug abuse, as determined by the Investigator.
* Current malignant disease (with the exception of basal cell carcinoma; BCC).
* Any serious or active medical or psychiatric illness, which in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol.
* Patients not willing/able to follow the study instructions.
* Resistance to aztreonam, or intolerance to aztreonam or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in Burkholderia spp. density in expectorated sputum and/or induced sputum. | 28 days, i.e. at start and end of treatment

SECONDARY OUTCOMES:
Clinical safety as measured by vital signs | Time Frame: Screening, day 0, 14, 28, 56, 70, 84 and follow up at day 112
  Measurement of vital signs
Clinical safety as measured by ECG | Time Frame: Screening, day 0, 14, 28, 56, 70, 84 and follow upat day 112
  Measurement of ECG
Clinical safety as measured by blood oxygen saturation | Time Frame: Screening, day 0, 14, 28, 56, 70, 84 and follow upat day 112
  Measurement of blood oxygen saturation
Clinical safety as measured by FEV1 (Forced Expiratory Volume in 1 second) | Time Frame: Screening, day 0, 14, 28, 56, 70, 84 and follow up at day 112
  Measurement of pulmonary function tests

CONTACTS AND LOCATIONS:
Overall Officials: Rainald Fischer, MD, PD, Principal Investigator — Pneumologische Praxis Pasing
Locations (2):
- Germany (2):
  - Pneumologische Praxis Pasing, Münich, Münich-Pasing
  - Charité Universitätsmedizin Berlin, Berlin

REFERENCES:
- [Derived] Fischer R, Schwarz C, Weiser R, Mahenthiralingam E, Smerud K, Meland N, Flaten H, Rye PD. Evaluating the alginate oligosaccharide (OligoG) as a therapy for Burkholderia cepacia complex cystic fibrosis lung infection. J Cyst Fibros. 2022 Sep;21(5):821-829. doi: 10.1016/j.jcf.2022.01.003. Epub 2022 Jan 24. PMID 35086790
- [Derived] Hurley MN, Smith S, Forrester DL, Smyth AR. Antibiotic adjuvant therapy for pulmonary infection in cystic fibrosis. Cochrane Database Syst Rev. 2020 Jul 16;7(7):CD008037. doi: 10.1002/14651858.CD008037.pub4. PMID 32671834